CLINICAL TRIAL: NCT00141011
Title: ASP I (Ancrod Stroke Program) Study of Acute Viprinex™ for Emergency Stroke: A Randomized, Double-Blind, Placebo-Controlled Study of Ancrod (Viprinex™) in Subjects Beginning Treatment Within 6 Hours of the Onset of Acute, Ischemic Stroke
Brief Title: Ancrod (Viprinex™) for the Treatment of Acute, Ischemic Stroke
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility
Sponsor: Neurobiological Technologies (Industry)
Responsible Party: Warren W. Wasiewski, M.D., Neurobiological Technologies, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTI-ASP-0502
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Stroke; Cerebral Ischemia; Brain Infarction
Keywords: Stroke; Fibrinogen; Reperfusion; Thrombolysis
MeSH Terms: conditions — Stroke; Brain Ischemia; Brain Infarction | interventions — Ancrod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous ancrod (Experimental): Intravenous ancrod infused at a rate of 0.167 IU/kg/hr (0.6 mL/kg/hr) for 2 or 3 hours depending on the pretreatment fibrinogen level.
  Interventions: Drug: Ancrod (Viprinex)
- Intravenous Placebo (Placebo Comparator): Intravenous placebo at a rate of 0.6 mL/kg/hr for 2 or 3 hours depending on the pretreatment fibrinogen level.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ancrod (Viprinex) — 0.167 IU/kg/hr (0.6 mL/kg/hr) IV for 2-3 hours
  Arms: Intravenous ancrod
Drug: Placebo — 0.6 mL/kg/hr
  Arms: Intravenous Placebo

SUMMARY:
The primary purpose of this study is to determine whether a brief intravenous infusion of ancrod started within 6 hours of stroke onset improves functional outcome at 3 months.

DETAILED DESCRIPTION:
With prior approval by the FDA, an interim analysis for futility was performed when 500 subjects had been entered into the two parallel trials, NCT00141001 and NCT00300196. The analyses were reviewed by the data safety monitoring board, which recommended that both studies be terminated because of futility. This was done at a point where 650 subjects had been entered into both studies, combined, but analyses were conducted only on the initial 500 subjects. Results of the abbreviated analysis will be found with study NCT00141001 since that study contributed most of the subjects to the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Acute, ischemic stroke with first symptoms within 6 hours of beginning treatment
* Baseline NIHSS > 5

Exclusion Criteria:

* No intracranial, extravascular blood on CT
* Hypertension (systolic > 185; diastolic > 105)
* Baseline fibrinogen level < 100 mg/dL
* Thrombocytopenia (< 100,000 / mm3)
* Recent (< 3 days) or anticipated (< 5 days) use of a thrombolytic agent
* Recent (< 14 days) or anticipated surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2005-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Responder analysis based on Modified Rankin Scale (mRS) | 90 days

SECONDARY OUTCOMES:
National Institute of Health Stroke Scale (NIHSS),Barthel Index (BI),Fibrinogen levels with ancrod tx, and Safety of ancrod tx | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Warren Wasiewski, M.D., Study Director — Neurobiological Technologies
Locations (100):
- United States (58):
  - Mayo Clinic Hospital / Arizona, Phoenix, Arizona
  - Sparks Regional Medical Center, Fort Smith, Arkansas
  - Loma Linda University School of Medicine, Loma Linda, California
  - Santa Monica - UCLA Medical Center, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Hoag Memorial Hospital, Newport Beach, California
  - The Neurology Center: Tri-City Medical Center, Oceanside, California
  - Shasta Regional Medical, Redding, California
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Neurologic Consultants, P.A., Fort Lauderdale, Florida
  - Shands Jacksonville / University of Florida, Jacksonville, Florida
  - Ocala Neurodiagnostic Center, Ocala, Florida
  - Florida Hospital Neuroloscience Institute, Orlando, Florida
  - Fawcett Memorial Hospital, Port Charlotte, Florida
  - Peace River Regional Medical Center, Port Charlotte, Florida
  - Tallahassee Memorial Healthcare, Inc., Tallahassee, Florida
  - The Queens Medical Center, Neuroscience Institute, Honolulu, Hawaii
  - Mercy Hospital, Chicago, Illinois
  - Elkhart Clinic, LLC - Neurology, Elkhart, Indiana
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Parkview Research Center, Fort Wayne, Indiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - Wayne State University, Detroit, Michigan
  - St. Mary's Duluth Clinic, Duluth, Minnesota
  - Minneapolis Clinic of Neurology, Golden Valley, Minnesota
  - Deaconess Billings Clinical Research Center, Billings, Montana
  - NJ Neuroscience Institute, Edison, New Jersey
  - Neurology Consultants Of Burlington County, Lumberton, New Jersey
  - UMDNJ / Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Neurology Group of Bergen County, Ridgewood, New Jersey
  - Shore Neurology, Toms River, New Jersey
  - Kaleida Stroke Center, Buffalo, New York
  - United Health Services Hospitals, Johnson City, New York
  - Winthrop University Hospital, Minneola, New York
  - Weill Medical College of Cornell University, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Strong Memorial Hospital, Rochester, New York
  - Presbyterian Hospital, Charlotte, North Carolina
  - Lebauer Cardiovascular Research Foundation at Moses Cone Hospital, Greensboro, North Carolina
  - Clinical Research of Winston-Salem, Winston-Salem, North Carolina
  - The Toledo Hospital, Toledo, Ohio
  - Medical University of Ohio, Toledo, Ohio
  - Northshore Clinical Associates, Erie, Pennsylvania
  - Westmoreland Neurology Associates, Inc., Greensburg, Pennsylvania
  - Miriam Hospital, Providence, Rhode Island
  - Beaufort Memorial Hospital, Beaufort, South Carolina
  - Methodist University Hospital, Memphis, Tennessee
  - Brackenridge Hospital, Austin, Texas
  - Seton Medical Center, Austin, Texas
  - Methodist Hospital / Neurological Institute, Houston, Texas
  - University of Texas Health Sciences Center, San Antonio, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Neurological Consultants of Virginia Beach, Virginia Beach, Virginia
  - Harborview Medical Center, Seattle, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - St. Lukes Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - Gosford Hospital Department of Neurology, Gosford, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - National Stroke Research Institute, Heidelberg Heights, Victoria
- Canada (7):
  - Grey Nuns Community Hospital, Edmonton, Alberta
  - Western Memorial Health Clinic, Corner Brook, Newfoundland and Labrador
  - London Health Sciences Centre - University Hospital, London, Ontario
  - Trillum Health Centre, Mississauga, Ontario
  - Hospital Charles-Leymoyne, Greenfield Park, Quebec
  - University of Alberta Hospital, Edmonton
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay
- Czechia (2):
  - St. Anne's Faculty Hospital, Brno
  - Faculty Hospital 1, The Clinic of Neurology, Pilsen
- St. Anna Hospital, Geldrop, Netherlands
- University Clinical Hospital, Warsaw, Poland
- Russia (3):
  - City Hospital #31, Moscow
  - Research Institute of Neurology RAMS, Moscow
  - Military Medical Akademy Dept of Neurology, Saint Petersburg
- South Africa (4):
  - St. Augustine's Hospital, Berea, Durban, KwaZulu-Natal
  - Tiervlei Trial Centre, Cape Town
  - Vergelegen Medi-Clinic, Somerset West
  - Sunninghill Hospital, Sunninghill
- Taiwan (17):
  - Changhua Christian Hospital, Chief Department of Neurology, Changhua
  - Lo-Tung Pohai Hospital, Department of Neurology, IIan
  - Chung-Ho Memorial Hospital Kaohsiung Medical University, Kaohsiung City
  - Kaohsiung Chang-Gung, Memorial Hospital, Kaohsiung City
  - Chung Shan Medical Hospital, Taichung
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Section of Neurology, Taichung
  - Kuang-Tien General Hospital, Taichung
  - Chi-Mei Medical Center, Tainan
  - National Taiwan University Hospital, Taipei
  - Cathay General Hospital Department of Neurology, Taipei
  - Shin-Kong WHS Memorial Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Far Eastern Memorial Hospital, Taipei
  - En Chu Kong Hospital, Taipei
  - Chang-Gung Memorial Hospital Linko Medical Center, Taoyuang
  - Chang-Gung Memorial Hospital, Linko Medical Center, Taoyuang
- United Kingdom (3):
  - University of Aberdeen, Polwarth Building, Institute of Medical Sciences, Dept. of Medicine & Theropeutics, Aberdeen
  - Institute of Neurological Sciences Southern General Hospital, Glasgow
  - Royal Victoria Infirmary - Clinical Research Center, Newcastle

REFERENCES:
- See also: Related Info — http://www.ntii.com